CLINICAL TRIAL: NCT05431270
Title: A Phase 1, Open-Label, Dose Escalation and Expansion Study of Mavrostobart (PT199) Administered Alone in Adult Patients with Advanced Solid TuMORs, in CombiNation with a Checkpoint INhibitor TreatinG Wild-type Non-Small Cell Lung Cancer, or in Combination with ChemoTherapy for Metastatic or Advanced PAncreatic Ductal AdenocaRcinoma (MORNINGSTAR)
Brief Title: Dose Escalation/Expansion Study of Mavrostobart (PT199), an Anti-CD73 MAb, Administered Alone and in Combination with a PD-1 Inhibitor or Chemotherapy (the MORNINGSTAR Study)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Phanes Therapeutics (Industry)
Collaborators: BeiGene (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PT199X1101
Record Dates: First submitted 2022-05-25; First posted 2022-06-24 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Non Small Cell Lung Cancer; Pancreatic Ductal Adenocarcinoma
Keywords: Advanced; Metastatic; Refractory; Anti-CD73; Checkpoint immunotherapies; PD-1/PD-L1 inhibitors
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasm Metastasis | interventions — tislelizumab; Gemcitabine; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; Docetaxel; Pemetrexed; Carboplatin; pembrolizumab

STUDY DESIGN:
Intervention Model Description: The study will consist of 4 parts: Monotherapy Dose Escalation (Part A), ICI Combination Therapy Dose Escalation (Part B), ICI Combination Dose Expansion in NSCLC (Part C), and Combination with Chemotherapy in frontline (1L) PDAC patients (Part D).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Part A: Monotherapy Dose Escalation (Experimental): A standard 3+3 dose escalation design will be employed, and 3 patients will be enrolled initially at each dose level. Mavrostobart (PT199) will be administered as a monotherapy.
  Interventions: Drug: Mavrostobart (PT199)
- Part B: Combination Therapy Dose Escalation (Experimental): A standard 3+3 dose escalation design will be employed, and 3 patients will be enrolled initially at each dose level. Patients will be treated with Mavrostobart (PT199) in combination with a PD-1 inhibitor, tislelizumab.
  Interventions: Drug: Mavrostobart (PT199); Drug: Tislelizumab
- Part C: Combination Therapy Dose Expansion (Experimental): Two RDEs for Part C will be determined in Part B and will be further evaluated in two dose expansion cohorts. Patients will be treated with Mavrostobart (PT199) in combination with a PD-1 inhibitor, tislelizumab.
  Interventions: Drug: Mavrostobart (PT199); Drug: Tislelizumab
- Part D: Chemotherapy Combination (Experimental): The Chemotherapy Combination Therapy Dose Escalation and Expansion will investigate four cohorts, one in frontline PDAC, two in frontline NSCLC and one in second-line and later NSCLC patients. Patients will receive Mavrostobart (PT199) plus chemotherapy, with one cohort also receiving pembrolizumab.
  Interventions: Drug: Mavrostobart (PT199); Drug: Gemcitabine + nab-Paclitaxel; Drug: Docetaxel; Drug: Pemetrexed; Drug: Gemcitabine; Drug: Carboplatin + Pemetrexed; Drug: Pembrolizumab + Carboplatin + Pemetrexed

INTERVENTIONS:
Drug: Mavrostobart (PT199) — Mavrostobart (PT199) is an anti-CD73 mAb with a differentiated mechanism of action.
Drug: Tislelizumab — Anti-PD-1 monoclonal antibody 200 mg Q3W, inhibits the lymphocytes PD-1 receptors, blocking the ligands that would deactivate it and prevent an immune response.
  Arms: Part B: Combination Therapy Dose Escalation; Part C: Combination Therapy Dose Expansion
Drug: Gemcitabine + nab-Paclitaxel — Dosing is per Standard of Care.
  Other Names: abraxane
  Arms: Part D: Chemotherapy Combination
Drug: Docetaxel — Dosing is per Standard of Care.
  Arms: Part D: Chemotherapy Combination
Drug: Pemetrexed — Dosing is per Standard of Care.
  Arms: Part D: Chemotherapy Combination
Drug: Gemcitabine — Dosing is per Standard of Care.
  Arms: Part D: Chemotherapy Combination
Drug: Carboplatin + Pemetrexed — Dosing is per Standard of Care.
  Arms: Part D: Chemotherapy Combination
Drug: Pembrolizumab + Carboplatin + Pemetrexed — Dosing is per Standard of Care.
  Arms: Part D: Chemotherapy Combination

SUMMARY:
This is a first-in-human, Phase 1/2, open-label, study designed to evaluate the safety, tolerability, pharmacokinetics, pharmacodynamics, and preliminary efficacy of Mavrostobart (PT199) alone and in combination with a PD-1 inhibitor or chemotherapy.

DETAILED DESCRIPTION:
Mavrostobart (PT199) is an anti-CD73 mAb with a differentiated mechanism of action and is expected to completely inhibit CD73 enzyme activity. Mavrostobart (PT199) is designed to counter the adenosine-mediated immunosuppressive tumor microenvironment, rendering anti-tumor immune cells to be more active and more responsive to checkpoint immunotherapies, such as PD-1/PD-L1 inhibitors.

CD73 is widely overexpressed in a number of different cancers, including pancreatic ductal adenocarcinoma (PDAC), gastric carcinoma, colorectal carcinoma, non-small cell lung cancer (NSCLC), sarcomas and glioblastomas. Thus, targeting CD73 may provide benefit for patients with a high CD73 expression in their tumor.

Mavrostobart (PT199) addresses the limitations of current CD73 inhibitors and is expected to increase antitumor immune activation, especially in combination with PD-1 pathway inhibition, and thus offer a new treatment option for cancer patients.

NSCLC is known to have a high expression level of CD73, and emerging clinical data has shown that targeting CD73 may provide clinical benefit, when combined with an immune checkpoint inhibitor (ICI) and/or standard of care chemotherapies to overcome treatment resistance.

ELIGIBILITY:
Key Inclusion Criteria

1. At least one measurable lesion as defined by RECIST V1.1 criteria for solid tumors.
2. For Part A: a histologically or cytologically confirmed unresectable advanced or metastatic solid tumors previously treated with therapies, or for which treatment is not available or not tolerated.

   For Part B: A histologically or cytologically confirmed diagnosis of NSCLC without actionable genomic alterations (AGAs) such as EGFR or ALK mutations and radiological documentation of disease progression on prior treatments, which may include a checkpoint inhibitor, or patients diagnosed with metastatic and/or advanced (m/a) PDAC who have disease progression after previously treated with therapies, or for which treatment is not available or not tolerated.

   For Part C: A histologically or cytologically confirmed diagnosis of NSCLC without actionable genomic alterations such as EGFR or ALK mutations and radiological documentation of disease progression on prior treatments, which may include a checkpoint inhibitor.

   For Part D:
   * Cohort D1: a histologically or cytologically confirmed diagnosis of pancreatic ductal adenocarcinoma (PDAC), treatment naïve for advanced or metastatic disease, and eligible to receive standard of care treatment with gemcitabine plus nab-paclitaxel.
   * Cohort D2: a histologically or cytologically confirmed diagnosis of NSCLC without actionable genomic alterations (AGAs) such as EGFR or ALK mutations and radiological documentation of disease progression on prior treatments, which may include a checkpoint inhibitor. Patients have progressed under first-line (1L) SOC chemotherapy with or without ICI or later lines of therapy, or for which standard 1L therapy has proven to be ineffective, intolerable, or is considered inappropriate.
   * Cohort D3: a histologically or cytologically confirmed diagnosis of NSCLC without actionable genomic alterations (AGAs) such as EGFR or ALK mutations. Patients are treatment naïve and have no contra indication to receive carboplatin plus pemetrexed.
   * Cohort D4: a histologically or cytologically confirmed diagnosis of NSCLC without actionable genomic alterations (AGAs) such as EGFR or ALK mutations. Patients are treatment naïve and are eligible for 1L therapy with pembrolizumab and carboplatin plus pemetrexed.
3. In all Parts, should be able to provide a tumor tissue sample (archival or newly acquired biopsy) to be assessed for CD73 and other biomarkers (PD-L1), unless deemed by the Investigator to cause risk to the patient or per Investigator's discretion.
4. ECOG performance status of 0 or 1.
5. Adequate organ function confirmed at screening and within 72 hours of initiating treatment.

Key Exclusion Criteria

1. Women who are pregnant or lactating.
2. Women of child-bearing potential (WOCBP) who do not use adequate birth control.
3. Autoimmune disease requiring systemic treatment within the past twelve months. Active autoimmune disease or a history of autoimmune diseases that may relapse.
4. Condition requiring systemic treatment with either corticosteroids or other immunosuppressive medications within 14 days prior to study treatment.
5. Patients who have experienced Grade ≥ 3 immune-related events, such as (non-infectious) pneumonitis, interstitial lung disease, myocarditis.
6. Patients with untreated brain or central nervous system (CNS) metastases or brain/CNS metastases that have progressed.
7. Impaired cardiac function or significant diseases.
8. Patients who have ≥ Grade 3 neuropathy.
9. Patients who have received wide field radiotherapy ≤ 4 weeks or limited field radiation for palliation ≤ 2 weeks prior to starting study drug or who have not recovered from adverse events of prior therapy.
10. Patients who are currently receiving (last dose within 5 days from C1D1) treatment with therapeutic doses of warfarin sodium (Coumadin®) or any other coumarin-derivative anticoagulants.

Additional inclusion and exclusion criteria will apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-08-11 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
To determine the maximum tolerated dose (MTD), if reached. | Start of the study drug till 90 days after last dose.
Recommended Phase 2 Dose of Mavrostobart (PT199) as a single agent and/or in combination with a PD-1 inhibitor. | Start of the study drug till 90 days after last dose.
Dose Limiting Toxicity (DLT). | Time Frame: Start of the study drug till 90 days after last dose.

SECONDARY OUTCOMES:
Preliminary efficacy assessed by the response rate by RECIST 1.1 for overall response rate. | Start of the study drug till 90 days after last dose.
Area Under the Curve from time 0 to last (AUC0-last) of Mavrostobart (PT199) | Time Frame: Start of the study drug till 90 days after last dose.
Maximum Concentration (Cmax) of Mavrostobart (PT199) | Time Frame: Start of the study drug till 90 days after last dose.
Half Life (T1/2) of Mavrostobart (PT199) | Time Frame: Start of the study drug till 90 days after last dose.
Preliminary efficacy assessed by the response rate by RECIST 1.1 for disease control rate. | Time Frame: Start of the study drug till 90 days after last dose.
Progression free survival duration. | Time Frame: Start of the study drug till 90 days after last dose.
6-month overall survival. | Time Frame: Start of the study drug till 90 days after last dose.

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Carolina BioOncology Institute, Huntersville, North Carolina
  - Sarah Cannon Research Institute University of Oklahoma, Oklahoma City, Oklahoma
  - SCRI Oncology Partners, Nashville, Tennessee
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Tranquility Research, Webster, Texas
  - NEXT Oncology, Fairfax, Virginia